CLINICAL TRIAL: NCT02672423
Title: A Bioequivalence Study Comparing Abemaciclib Capsule and Tablet Formulations and Effect of Food on Abemaciclib Tablet Pharmacokinetics in Healthy Subjects
Brief Title: A Study of Abemaciclib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16169; I3Y-MC-JPCC (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abemaciclib Part A (Experimental): Reference formulation (R) = 3 x 50 mg abemaciclib capsules, Test formulation (T150) = 150 mg abemaciclib tablet administered orally on Day 1 in each of 2 periods.
  Interventions: Drug: Abemaciclib Capsules (Reference Formulation); Drug: Abemaciclib Tablet (Test Formulation)
- Abemaciclib Part B (Experimental): R = 3 x 50 mg abemaciclib capsules, T150 = 150 mg abemaciclib tablet, Test Formulation 50 (T50) = 3 x 50 mg abemaciclib tablets administered orally on Day 1 in each of 3 periods.
  Interventions: Drug: Abemaciclib Capsules (Reference Formulation); Drug: Abemaciclib Tablet (Test Formulation)
- Abemaciclib Part C (Experimental): T150 Fed and T150 Fasted = 150 mg abemaciclib tablet with a high-fat meal (T150 Fed) and then without a high-fat meal (T150 Fasted) on Day 1 in each of 2 periods administered orally.
  Interventions: Drug: Abemaciclib Tablet (Test Formulation)

INTERVENTIONS:
Drug: Abemaciclib Capsules (Reference Formulation) — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib Part A; Abemaciclib Part B
Drug: Abemaciclib Tablet (Test Formulation) — Administered orally
  Other Names: LY2835219

SUMMARY:
The purpose of this study is to measure how much abemaciclib gets into the blood stream and how long it takes the body to get rid of it when given as capsules versus a tablet(s). The effect of a high fat meal on the tablet formulation will also be evaluated. In addition, the tolerability of abemaciclib tablet and capsule formulations will be evaluated. Information about any side effects that may occur will also be collected.

This study has 3 parts. Parts A and C will last about 44 days including follow-up. Part B will last about 60 days including follow-up. Screening may occur up to 28 days before the first dose of study drug. Participants are only allowed to enroll in one part.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy surgically sterile or postmenopausal females and sterile males
* Have a body mass index (BMI) 18 to 32 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Have known allergies to abemaciclib, related compounds, or any components of the formulation
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Daytona Beach Clinical Research Unit, Daytona Beach, Florida
  - Evansville Clinical Research Unit, Evansville, Indiana

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 2- and 3-period crossover study conducted in 3 parts, with Part A followed by Parts B and C. Participants received single oral doses of abemaciclib on 2 separate occasions in Parts A and C and on 3 separate occasions in Part B.There was a washout interval of at least 16 days between periods.
Groups:
- Part A: Abemaciclib (R,T150 ): Reference formulation (R) = 3 x 50 mg abemaciclib capsules, Test formulation (T150) = 150 mg abemaciclib tablet administered orally on Day 1 in each of 2 periods.
- Part A: Abemaciclib (T150,R): T150 = 150 mg abemaciclib tablet, R = 3 x 50 mg abemaciclib capsules administered orally on Day 1 in each of 2 periods.
- Part B: Abemaciclib (R,T150,T50 ): R = 3 x 50 mg abemaciclib capsules, T150 = 150 mg abemaciclib tablet, Test Formulation 50 (T50) = 3 x 50 mg abemaciclib tablets administered orally on Day 1 in each of 3 periods.
- Part B: Abemaciclib (T150,T50,R); Part B: Abemaciclib (T150,R,T50): T150 = 150 mg abemaciclib tablet, R = 3 x 50 mg abemaciclib capsules, T50 = 3 x 50 mg abemaciclib tablets administered orally on Day 1 in each of 3 periods.
- Part B: Abemaciclib (T50,R,T150): T50 = 3 x 50 mg abemaciclib tablets, R = 3 x 50 mg abemaciclib capsules, T150 = 150 mg abemaciclib tablet administered orally on Day 1 in each of 3 periods.
- Part B: Abemaciclib (R,T50,T150): R = 3 x 50 mg abemaciclib capsules, T50 = 3 x 50 mg abemaciclib tablets, T150 = 150 mg abemaciclib tablet administered orally on Day 1 in each of 3 periods.
- Part B: Abemaciclib (T50,T150,R): T50 = 3 x 50 mg abemaciclib tablets, T150 = 150 mg abemaciclib tablet, R = 3 x 50 mg abemaciclib capsules administered orally on Day 1 in each of 3 periods.
- Part C: Abemaciclib (T150 Fed, T150 Fasted): T150 Fed and T150 Fasted = 150 mg abemaciclib tablet with a high-fat meal (T150 Fed) and then without a high-fat meal (T150 Fasted) on Day 1 in each of 2 periods administered orally.
- Part C: Abemaciclib (T150 Fasted, T150 Fed): T150 Fasted and T150 Fed = 150 mg abemaciclib tablet with a high-fat meal (T150 Fed) and then without a high-fat meal (T150 Fasted) on Day 1 in each of 2 periods administered orally.
Period: Period 1
Arm/Group | Part A: Abemaciclib (R,T150 ) | Part A: Abemaciclib (T150,R) | Part B: Abemaciclib (R,T150,T50 ) | Part B: Abemaciclib (T150,T50,R) | Part B: Abemaciclib (T50,R,T150) | Part B: Abemaciclib (R,T50,T150) | Part B: Abemaciclib (T150,R,T50) | Part B: Abemaciclib (T50,T150,R) | Part C: Abemaciclib (T150 Fed, T150 Fasted) | Part C: Abemaciclib (T150 Fasted, T150 Fed)
Started | 7 | 7 | 14 | 15 | 15 | 15 | 15 | 15 | 12 | 12
Received at Least One Dose of Study Drug | 7 | 7 | 14 | 15 | 15 | 15 | 15 | 15 | 12 | 12
Completed | 7 | 7 | 14 | 15 | 14 | 15 | 15 | 15 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout 1
Arm/Group | Part A: Abemaciclib (R,T150 ) | Part A: Abemaciclib (T150,R) | Part B: Abemaciclib (R,T150,T50 ) | Part B: Abemaciclib (T150,T50,R) | Part B: Abemaciclib (T50,R,T150) | Part B: Abemaciclib (R,T50,T150) | Part B: Abemaciclib (T150,R,T50) | Part B: Abemaciclib (T50,T150,R) | Part C: Abemaciclib (T150 Fed, T150 Fasted) | Part C: Abemaciclib (T150 Fasted, T150 Fed)
Started | 7 | 7 | 14 | 15 | 14 | 15 | 15 | 15 | 12 | 12
Completed | 7 | 7 | 14 | 15 | 14 | 15 | 15 | 15 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part A: Abemaciclib (R,T150 ) | Part A: Abemaciclib (T150,R) | Part B: Abemaciclib (R,T150,T50 ) | Part B: Abemaciclib (T150,T50,R) | Part B: Abemaciclib (T50,R,T150) | Part B: Abemaciclib (R,T50,T150) | Part B: Abemaciclib (T150,R,T50) | Part B: Abemaciclib (T50,T150,R) | Part C: Abemaciclib (T150 Fed, T150 Fasted) | Part C: Abemaciclib (T150 Fasted, T150 Fed)
Started | 7 | 7 | 14 | 15 | 14 | 15 | 15 | 15 | 12 | 12
Completed | 7 | 7 | 13 | 15 | 14 | 15 | 15 | 15 | 12 | 12
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2
Arm/Group | Part A: Abemaciclib (R,T150 ) | Part A: Abemaciclib (T150,R) | Part B: Abemaciclib (R,T150,T50 ) | Part B: Abemaciclib (T150,T50,R) | Part B: Abemaciclib (T50,R,T150) | Part B: Abemaciclib (R,T50,T150) | Part B: Abemaciclib (T150,R,T50) | Part B: Abemaciclib (T50,T150,R) | Part C: Abemaciclib (T150 Fed, T150 Fasted) | Part C: Abemaciclib (T150 Fasted, T150 Fed)
Started | 7 | 7 | 13 | 15 | 14 | 15 | 15 | 15 | 12 | 12
Completed | 7 | 7 | 13 | 15 | 14 | 15 | 15 | 15 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A: Abemaciclib (R,T150 ) | Part A: Abemaciclib (T150,R) | Part B: Abemaciclib (R,T150,T50 ) | Part B: Abemaciclib (T150,T50,R) | Part B: Abemaciclib (T50,R,T150) | Part B: Abemaciclib (R,T50,T150) | Part B: Abemaciclib (T150,R,T50) | Part B: Abemaciclib (T50,T150,R) | Part C: Abemaciclib (T150 Fed, T150 Fasted) | Part C: Abemaciclib (T150 Fasted, T150 Fed)
Started | 0 (Part A was a 2-period study design.) | 0 (Part A was a 2-period study design.) | 13 | 15 | 14 | 15 | 15 | 15 | 0 (Part C was a 2-period study design.) | 0 (Part C was a 2-period study design.)
Completed | 0 | 0 | 13 | 15 | 14 | 14 | 15 | 14 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Part A: Abemaciclib: Reference formulation (R) = 3 x 50 mg abemaciclib capsules, Test formulation (T150) = 150 mg abemaciclib tablet administered orally on Day 1 in each of 2 periods.
- Part B Abemaciclib: R = 3 x 50 mg abemaciclib capsules, T150 = 150 mg abemaciclib tablet, Test Formulation 50 (T50) = 3 x 50 mg abemaciclib tablets administered orally on Day 1 in each of 3 periods.
- Part C Abemaciclib: T150 Fed and T150 Fasted = 150 mg abemaciclib tablet with a high-fat meal (T150 Fed) and then without a high-fat meal (T150 Fasted) on Day 1 in each of 2 periods administered orally.
- Total: Total of all reporting groups
Arm/Group | Part A: Abemaciclib | Part B Abemaciclib | Part C Abemaciclib | Total
Number analyzed (Participants) | 14 | 89 | 24 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (16.9) | 51.8 (11.6) | 55.5 (10.6) | 52.7 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 78 | 21 | 110
  Male | 3 | 11 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 24 | 10 | 38
  Not Hispanic or Latino | 10 | 65 | 14 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 13 | 0 | 16
  White | 9 | 69 | 22 | 100
  More than one race | 2 | 6 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 89 | 24 | 127

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞])
Description: Area under the concentration versus time curve from zero to infinity.
Time Frame: Parts A and C Periods 1 and 2; Part B Periods 1, 2, 3: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 96, 120,144,168 and 192 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour/milliliter (ng*hr/mL)
Groups:
- Part A: 150 mg Abemaciclib (T150); Part B: 150 mg Abemaciclib (T150): 150 mg abemaciclib tablet (test formulation[T150]) administered orally on Day 1 of 1 period.
- Part A: 3 x 50 mg Abemaciclib (R); Part B: 3 x 50 mg Abemaciclib (R): 3 x 50 mg abemaciclib capsules (reference formulation[R]) administered orally on Day 1 of 1 period.
- Part B: 3 x 50 mg Abemaciclib (T50): 3 x 50 mg abemaciclib tablets (T50) administered orally on Day 1 of 1 period.
- Part C: 150 mg Abemaciclib (Fed): 150 mg abemaciclib tablet (test formulation [T150]) with a meal administered orally on Day 1 of 1 period.
- Part C: 150 mg Abemaciclib (Fasted): 150 mg abemaciclib tablet (test formulation[T150]) without a meal administered orally on Day 1 of 1 period.
Arm/Group | Part A: 150 mg Abemaciclib (T150) | Part A: 3 x 50 mg Abemaciclib (R) | Part B: 150 mg Abemaciclib (T150) | Part B: 3 x 50 mg Abemaciclib (T50) | Part B: 3 x 50 mg Abemaciclib (R) | Part C: 150 mg Abemaciclib (Fed) | Part C: 150 mg Abemaciclib (Fasted)
Number analyzed (Participants) | 13 | 12 | 82 | 85 | 84 | 23 | 24
Nanograms*hour/milliliter (ng*hr/mL) | 3080 (57) | 2880 (56) | 3110 (55) | 3120 (52) | 3130 (59) | 4170 (49) | 3590 (45)

2. Primary Outcome: PK: Maximum Observed Drug Concentration (Cmax)
Description: Maximum observed drug concentration.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Groups:
- Part A: 3 x 50 mg Abemaciclib (R); Part B: 3 x 50 mg Abemaciclib (R): 3 x 50 mg abemaciclib capsules (reference formulation [R]) administered orally on Day 1 of 1 period.
- Part B:150 mg Abemaciclib (T150): 150 mg abemaciclib tablet (test formulation [T150]) administered orally on Day 1 of 1 period.
- Part C:150 mg Abemaciclib (Fed): 150 mg abemaciclib tablet (test formulation[T150]) with a meal administered orally on Day 1 of 1 period.
- Part C:150 mg Abemaciclib (Fasted): 150 mg abemaciclib tablet (test formulation[T150]) without a meal administered orally on Day 1 of 1 period.
Arm/Group | Part A: 150 mg Abemaciclib (T150) | Part A: 3 x 50 mg Abemaciclib (R) | Part B:150 mg Abemaciclib (T150) | Part B: 3 x 50 mg Abemaciclib (T50) | Part B: 3 x 50 mg Abemaciclib (R) | Part C:150 mg Abemaciclib (Fed) | Part C:150 mg Abemaciclib (Fasted)
Number analyzed (Participants) | 13 | 12 | 82 | 85 | 84 | 23 | 24
Nanograms per milliliter (ng/mL) | 104 (52) | 101 (56) | 95.2 (48) | 97.7 (50) | 95.8 (51) | 130 (44) | 99.6 (36)

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Part A: 3 x 50 mg (R): 3 x 50 milligrams (mg) abemaciclib capsules (reference formulation [R]) administered orally on Day 1 of 1 period.
- Part A: 1 x 150 mg (T150); Part B 1 x 150 mg (T150): 150 mg abemaciclib tablet (test formulation[T150]) administered orally on Day 1 of 1 period.
- Part B: 3 x 50 mg (R): 3 x 50 milligrams (mg) abemaciclib capsules (reference formulation[R]) administered orally on Day 1 of 1 period.
- Part B 3 x 50 mg (T50): 3 x 50 mg abemaciclib tablets (test formulation[T50]) administered orally on Day 1 of 1 period.
- Part C: (T150 Fed, T150 Fasted): 150 mg abemaciclib tablet (test formulation [T150]) with a meal and then without a meal administered orally on Day 1 of 1 period..
- Part C: (T150 Fasted, T150 Fed): 150 mg abemaciclib tablet (test formulation [T150]) without a meal and then with a meal administered orally on Day 1 of 1 period.
Arm/Group | Part A: 3 x 50 mg (R) | Part A: 1 x 150 mg (T150) | Part B: 3 x 50 mg (R) | Part B 1 x 150 mg (T150) | Part B 3 x 50 mg (T50) | Part C: (T150 Fed, T150 Fasted) | Part C: (T150 Fasted, T150 Fed)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/88 | 0/87 | 0/88 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 7/14 | 6/14 | 21/88 | 17/87 | 22/88 | 3/24 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 3 x 50 mg (R) (N=14) | Part A: 1 x 150 mg (T150) (N=14) | Part B: 3 x 50 mg (R) (N=88) | Part B 1 x 150 mg (T150) (N=87) | Part B 3 x 50 mg (T50) (N=88) | Part C: (T150 Fed, T150 Fasted) (N=24) | Part C: (T150 Fasted, T150 Fed) (N=24)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 5 (5) | 5 (5) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 8 (8) | 9 (9) | 12 (12) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 4 (5) | 5 (5) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 11 (11) | 7 (9) | 7 (7) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days